CLINICAL TRIAL: NCT02932215
Title: Pilot Study: Use of a Mobile Health Sensor in an Open Label Trial of Lorcaserin for the Treatment of Cannabis Use Disorder
Brief Title: Use of a Mobile Health Sensor in an Open Label Trial of Lorcaserin for the Treatment of Cannabis Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Christina Ann Brezing, research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7242
Record Dates: First submitted 2016-09-19; First posted 2016-10-13 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Cannabis Use Disorder
Keywords: mobile health device; substance abuse treatment; quality of life; lorcaserin
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental): All participants will receive open label lorcaserin
  Interventions: Drug: lorcaserin; Other: Fitbit Charge HR

INTERVENTIONS:
Drug: lorcaserin — Open label
  Other Names: Belviq
Other: Fitbit Charge HR — This is actually not an intervention- it is a tool to measure activity and sleep; all participants will be receiving one to collect data

SUMMARY:
This is a 10 week, open-label, prospective study, involving 10 volunteer participants with cannabis use disorder to test the feasibility and safety of using lorcaserin in addition to the feasibility, likability, and utility of a mobile sensor device in cannabis users. The study will be entirely outpatient. Upon study entry, participants will begin clinic visits at the Substance Treatment and Research Service (STARS) clinic. All consented participants will receive a Fitbit Charge HR device in week 1 to wear for the entire study and receive lorcaserin beginning in week 2 for a total of 8 weeks (weeks 2-9). At the beginning of week 10 following discontinuation of lorcaserin, the participants will continue to wear the Fitbit Charge HR device for this final week following completion of the medication trial. All participants will visit the clinic twice weekly to provide urine toxicology on THC, report on adverse events, complete additional assessments (outlined below), and upload de-identified data from the Fitbit Charge HR device to the secure encrypted Fitabase database. Study assessments will be collected at baseline, throughout the study, and 1 week following medication discontinuation. All participants will also receive medical management, a medication adherence focused psychosocial intervention that facilitates compliance with study medication and other study procedures, including adherence to wearing the Fitbit Charge HR device, and promotes abstinence from cannabis and other substances. Progressive voucher incentives will be provided for compliance with visit attendance and study procedures.

DETAILED DESCRIPTION:
Design Overview: This is a 10 week, open-label, prospective study, involving 10 volunteer participants with cannabis use disorder to test the feasibility and safety of using lorcaserin in addition to the feasibility, likability, and utility of a mobile sensor device in cannabis users. The study will be entirely outpatient Upon study entry, participants will begin clinic visits at the Substance Treatment and Research Service (STARS) clinic. All consented participants will receive a Fitbit charge HR mobile device in week 1 to wear for the entire study and receive lorcaserin beginning in week 2 for a total of 8 weeks (weeks 2-9). At the beginning of week 10 following discontinuation of lorcaserin, the participants will continue to wear the device for this final week following completion of the medication trial. All participants will visit the clinic twice weekly to provide urine toxicology on THC, report on adverse events, complete additional assessments (outlined below), and upload de-identified data from the device to a secure encrypted database. Study assessments will be collected at baseline, throughout the study, and 1 week following medication discontinuation. All participants will also receive medical management, a medication adherence focused psychosocial intervention that facilitates compliance with study medication and other study procedures, including adherence to wearing the device, and promotes abstinence from cannabis and other substances. Progressive voucher incentives will be provided for compliance with visit attendance and study procedures.

The specific aims of the project are:

1. To determine whether lorcaserin is associated with a reduction from baseline in cannabis use in individuals with cannabis use disorder seeking treatment.
2. To determine the tolerability of lorcaserin in this population.
3. To evaluate the feasibility and likability of incorporating a mobile health sensor device in a treatment study for cannabis use disorder.

The primary outcome measures are:

1. Lorcaserin will significantly reduce cannabis use during the study period as measured by self-report (Timeline Followback) and creatinine-normalized quantitative THC urine levels.
2. Lorcaserin will be well tolerated in participants with cannabis use disorder as measured by the proportion of participants completing the study, adherence to medication, and the proportion of participants experiencing adverse events.
3. Participants will find it feasible and likeable to utilize the Fitbit Charge HRTM in the study as measured by selfreport assessment of liking and adherence to wearing the device

Secondary aims include:

1. To evaluate the effect of medication treatment for cannabis use disorder on activity, sleep, stress, and quality of life as measured with a mobile sensor device and self-report assessments in individuals with cannabis use disorder.
2. To evaluate the correlation between summarized Fitbit Charge HR health sensor measures and self-report assessments of sleep, stress, and quality of life in addition to participants' use of cannabis and cannabis withdrawal at baseline, during, and after a treatment trial.

The secondary outcome measures include:

1. Medication treatment will increase positive health behaviors including activity and improve sleep (increase total sleep time and percentage deep sleep) in addition to decreasing stress and improving quality of life as measured by summarized daily total steps, sleep duration and quality, and summarized stress score measured with device in conjunction with improvement in the Pittsburgh Sleep Quality Inventory (PSQI), decreased Perceived Stress Scale score (PSS), and improvement on Quality of Life, Enjoyment, and Satisfaction Questionnaire (QLESQ), as compared to baseline. Negative health behaviors (poor sleep, decreased activity, increased stress) will be highest within subjects before starting treatment and with initial abstinence from cannabis when withdrawal symptoms are most prominent. Positive health behaviors will increase during treatment within subject, and particularly towards the second half of treatment as reduction in cannabis use or abstinence is sustained.
2. The device measures and self-report measures will directly correlate, as expected; ie: increased sleep and increased % of deep sleep will correlate with higher PSQI scores. When participants are using baseline levels of cannabis or are in cannabis withdrawal, they will have device measures consistent with negative health behaviors (poor sleep, decreased activity, increased stress). When they reduce cannabis use or achieve abstinence for a sustained period (any 14 days), an association with positive health behaviors as measured by the mobile device (adequate sleep, adequate activity, decreased stress) will increase.

The objective of the pilot is to obtain preliminary data on cannabis use patterns, tolerability of this medication, and sleep, quality of life and activity patterns in individuals with cannabis use disorder before conducting a larger trial with lorcaserin and to inform future applications of mobile sensors to cannabis use disorder treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-60
* Meets DSM-V criteria for a current cannabis use disorder
* Seeking treatment for cannabis use disorder
* THC-positive urine drug screen
* Capable of giving informed consent and complying with study procedures
* Has access to a mobile device with IOS7 or Android 4.4.2 capabilities or more recent operating systems
* Not underweight (Defined as BMI ≥18.5)

Exclusion Criteria:

* Lifetime history of DSM-V diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
* Current DSM-V criteria for any other psychiatric disorder supported by the MINI that in the investigator's judgment is unstable, would be disrupted by the study medication, or is likely to require new pharmacotherapy or psychotherapy during the study period. Individuals who are currently stable on a psychotropic medication for at least 3 months may be included if in the investigator's opinion the psychotropic medication the patient is taking is compatible with the study medication (lorcaserin).
* Individuals who meet DSM-V criteria for any substance use disorder other an cannabis, caffeine or nicotine use disorders
* Pregnancy, lactation, or failure to use adequate contraceptive method in female patients who are currently engaging in sexual activity with men
* Unstable medical conditions, such as AIDS, cancer, uncontrolled hypertension (blood pressure > 140/90), uncontrolled diabetes, pulmonary hypertension or heart disease
* Legally mandated to participate in a substance use disorder treatment program
* Current or recent history of significant violent orsuicidal behavior, risk for suicide or homicide psychiatrist
* Currently meets DSM-V diagnosis for an eating disorder or is underweight (defined as BMI <18.5)
* Elevated liver function tests (AST and ALT > 3 times the upper limit of normal) or impaired renal function
* Known history of allergy, intolerance, or hypersensitivity to lorcaserin
* Concurrent use of migraine medications ergotamine (Cafergot, Ergomar) or dihydroergotamine (Migranal), 5HT2B receptor agonists like cabergoline, or medications metabolized by CYP2D6 (thioridazine, tamoxifen, metoprolol, aripiprazole, codeine, etc)
* No access to mobile device with IOS7 or Android 4.4.2 capabilities or more recent operating systems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Cannabis use | weeks 1-10
  urine toxicology
Adherence to device | weeks 1-10
  days device is worn
Feasibility of implementing mobile health device in treatment trial for CUD | assessed once at 10weeks (end of study)
  5 question self-report on likability of device; eg: Question 1: did you like wearing the mobile sensor device to track your progress during treatment? Yes or No; Question 2: Would you continue to wear the mobile sensor device to track your behaviors? Yes or No; etc
Cannabis Use | weeks 1-10
  Timeline Followback
adherence to medication | weeks 1- 8
  number of pills taken

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia Substance Treatment and Research Service, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brezing CA, Sibai M, Choi CJ, Mitra S, Mariani JJ, Naqvi N, Mahony AL, Brooks D, Pavlicova M, Levin FR. Open Label Pilot of Lorcaserin (a serotonin 2C-receptor agonist) for Cannabis Use Disorder. J Subst Use. 2024;29(4):487-494. doi: 10.1080/14659891.2023.2202760. Epub 2023 May 10. PMID 39021751